CLINICAL TRIAL: NCT04040322
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Phase 3 Study Evaluating the Safety and Efficacy of Intravenous Iloprost in Subjects With Systemic Sclerosis Experiencing Symptomatic Digital Ischemic Episodes (AURORA Study)
Brief Title: Intravenous Iloprost in Subjects With Symptomatic Raynaud's Phenomenon Secondary to Systemic Sclerosis (Phase 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Civi Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ES-301
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Raynaud's Phenomenon Secondary to Systemic Sclerosis
Keywords: systemic sclerosis; raynaud's phenomenon
MeSH Terms: conditions — Scleroderma, Systemic; Raynaud Disease | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line. Study drug will be initiated at a starting dose 0.5 ng/kg/min up to 2.0 ng/kg/min.
  Interventions: Drug: Placebo IV infusion
- Iloprost Injection, for intravenous use (Active Comparator): Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line. Study drug will be initiated at a starting dose 0.5 ng/kg/min up to 2.0 ng/kg/min.
  Interventions: Drug: Iloprost Injection, for intravenous use

INTERVENTIONS:
Drug: Placebo IV infusion — Study drug will be initiated at a starting dose of 0.5 ng/kg/min up to 2.0 ng/kg/min. Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line.
  Arms: Placebo
Drug: Iloprost Injection, for intravenous use — Study drug will be initiated at a starting dose of 0.5 ng/kg/min up to 2.0 ng/kg/min. Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line.
  Arms: Iloprost Injection, for intravenous use

SUMMARY:
This is a Phase 3, multicenter, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of iloprost on the frequency of and relief from symptomatic digital ischemic episodes in subjects with systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects must be greater than or equal to 18 years of age.
* Subjects must have a diagnosis of Systemic Sclerosis as defined by the 2013 American College of Rheumatology criteria/EULAR criteria
* Subjects must have a diagnosis or history of Raynaud's Phenomenon, self-reported or reported by a physician, with at least a 2-phase color change in finger(s) of pallor, cyanosis, and/or reactive hyperemia in response to cold exposure or emotion
* Subjects must have a minimum of 10 symptomatic Raynaud's Phenomenon attacks, documented in the electronic patient-reported outcomes (ePRO) diary, occurring over at least 3 separate days of the 3- to 5-day eligibility period
* Subjects must complete a minimum of 80% of the daily ePRO diary entry during the baseline period
* Female subjects of childbearing potential and male subjects must agree to use contraception for the duration of the study.
* Subjects must be willing and able to comply with the study requirements and give informed consent for participation in the study

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding
* Subjects with systolic blood pressure <85 mmHg
* Subjects with an estimated glomerular filtration rate <15 mL/min/1.73 m2
* Subjects with an alanine aminotransferase and/or aspartate aminotransferase value >3 × the upper limit of normal at screening
* Subjects who have a digital ulcer infection within 30 days of screening
* Subjects with a history of cervical or digital sympathectomy, or botulism toxin injections in their hands [for RP or digital ulcers] within 90 days of screening. Subjects should not have a planned botulism toxin or sympathectomy during their participation in the study.
* Subjects with gangrene or digital amputation within 6 months of screening
* Subjects with current intractable diarrhea or vomiting
* Subjects with a risk of clinically significant bleeding events, including those with coagulation or platelet disorders at screening
* Subjects with a history of major trauma or hemorrhage within 30 days of screening.
* Subjects with clinically significant chronic intermittent bleeding, such as active gastric antral vascular ectasia or active peptic ulcer disease, within 60 days of screening
* Subjects who have had any cerebrovascular events (eg, transient ischemic attack or stroke) within 6 months of screening
* Subjects with a history of myocardial infarction or unstable angina within 6 months of screening. Subjects should not have a planned coronary procedure during their participation in the study
* Subjects with acute or chronic congestive heart failure (New York Heart Association Class III [moderate] or Class IV [severe]) at screening
* Subjects with a history of more than mild restrictive or congestive cardiomyopathy uncontrolled by medication or implanted device
* Subjects with a history of life-threatening cardiac arrhythmias
* Subjects with a history of hemodynamically significant aortic or mitral valve disease
* Subjects with a history of known pulmonary hypertension, pulmonary arterial hypertension, or pulmonary veno-occlusive disease
* Subjects with a history of significant restrictive lung disease, defined as forced vital capacity <45% predicted and diffusing capacity of the lungs for carbon monoxide <40% predicted (uncorrected for hemoglobin)
* Subjects with scleroderma renal crisis within 6 months of screening
* Subjects with a concomitant life-threatening disease with a life expectancy <12 months
* Subjects who have a clinically significant disorder that, in the opinion of the Investigator, could contraindicate the administration of study drug, affect compliance, interfere with study evaluations, or confound the interpretation of study results
* Subjects who have taken or are currently taking any parenteral, inhaled, or oral prostacyclin or prostacyclin receptor agonists (eg, epoprostenol, treprostinil, iloprost, and selexipag) within 8 weeks of screening
* Subjects who have initiated or had a dose change of any of the following within 2 weeks of screening: oral, topical, or intravenous (IV) vasodilators (eg, calcium channel blockers, phosphodiesterase-5 (PDE5) inhibitors [eg, sildenafil, tadalafil, or vardenafil], nitrates, and fluoxetine)
* Subjects with any history of acetaminophen intolerability (eg, allergic reaction to acetaminophen)
* Subjects with any malignancy that requires treatment during the study period, that has required treatment within 1 year of screening (including excision of skin cancer) or that is currently not in remission
* Subjects who have used any investigational medication or device for any indication within 30 days or 5 half-lives (whichever is longer)
* Subjects who have participated in ES-201 or ES-301 studies and were randomized and treated with study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Benton, Pharm D, Study Director — Eicos Sciences, Inc.
Locations (30):
- United States (30):
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - University of Arizona - Arthritis Research Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Georgetown University Medical Center - Department of Rheumatology, Washington D.C., District of Columbia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - West Michigan Rheumatology PLLC, Grand Rapids, Michigan
  - University of Minnesota Maple Grove, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati - Scleroderma Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - The University of Toledo Medical Center (UTMC) - Ruppert Health Center, Toledo, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - University of Texas Houston - Division of Rheumatology and Clinical Immunogenetics, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated on 14 October 2019 and completed on 07 May 2021. It was conducted in 31 sites located in the United States.
Pre-assignment Details: In this study 258 participants with Systemic Sclerosis (SSc) were screened.198 participants who had at least 10 symptomatic Raynaud's phenomenon (RP) attacks on the 5-day eligibility period were randomized: 98 to the placebo arm and 100 to the Iloprost arm. Two participants stopped the study prior to receiving any treatment. The number of participants who were randomized and started the treatment was 97 in the placebo arm and 99 in the Iloprost arm.
Groups:
- Placebo: Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line. Study drug will be initiated at a starting dose 0.5 ng/kg/min up to 2.0 ng/kg/min.
  Placebo IV infusion: Study drug will be initiated at a starting dose of 0.5 ng/kg/min up to 2.0 ng/kg/min.
  Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line.
- Iloprost Injection, for Intravenous Use: Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line. Study drug will be initiated at a starting dose 0.5 ng/kg/min up to 2.0 ng/kg/min.
  Iloprost Injection, for intravenous use: Study drug will be initiated at a starting dose of 0.5 ng/kg/min up to 2.0 ng/kg/min.
  Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line.
Period: Overall Study
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
Started | 97 | 99
Completed | 97 | 99
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use | Total
Number analyzed (Participants) | 97 | 99 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (10.92) | 52.4 (13.59) | 52.2 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 88 | 174
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 86 | 85 | 171
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 6 | 15
  White | 80 | 87 | 167
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Phosphodiesterase-5 (PDE5) Inhibitors at Screening [Count of Participants; unit: Participants]
  Yes | 37 | 40 | 77
  No | 60 | 59 | 119
Weekly frequency of symptomatic RP attacks at baseline [Mean (Standard Deviation); unit: Weekly frequency of RP attacks] | 28.63 (18.113) | 32.49 (26.393) | 30.58 (22.701)

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Symptomatic RP Attacks
Description: The primary efficacy parameter is the change in the weekly frequency of symptomatic RP attacks from baseline.
  The baseline weekly frequency of symptomatic RP attacks was defined as the average number of weekly symptomatic RP attacks that occurred during the 10- to 25-day baseline ePRO diary completion period.
  The double-blind endpoint weekly frequency of symptomatic RP attacks was defined as the average number of weekly symptomatic RP attacks that occurred during Days 8 to 21, inclusive
Time Frame: From baseline (Day 10 to Day 25 of screening period) to the end ofthe efficacy follow-up (Day 8 to Day 21).
Population: The Intention-To-Treat (ITT) Population was defined as all randomized patients who initiated (received) study drug infusion.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of RP attacks per week
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
Number analyzed (Participants) | 97 | 99
Number of RP attacks per week | -11.47 [-13.69 to -9.25] | -12.73 [-14.92 to -10.55]
Statistical Analysis 1: Comparison: Placebo vs Iloprost Injection, for Intravenous Use; Test type: Superiority; p = 0.4210, ANCOVA — Threshold for statistical significance was p < 0.05; Least squares mean difference in change = -1.26, 95% CI 2-sided [-4.34 to 1.82]

2. Secondary Outcome: Change in Severity of RP Attack Symptoms
Description: Change in overall severity of RP attack symptoms as registered in electronic diary. It was measured using an 11-point numeric rating scale (NRS) as follows: 0 = no pain/numbness/tingling/discomfort, 1 to 3 = mild pain/numbness/tingling/discomfort, 4 to 6 = moderate pain/numbness/tingling/discomfort, and 7 to 10 = severe pain/numbness/tingling/discomfort. The severity of the symptoms (pain, numbness, discomfort or tingling) was rated by the patient in the electronic diary (ePRO). The symptom with the worst average baseline value for each patient was compared to the average severity rate of that symptom which occurred during Days 8 to 21 of the treatment period. If more than 1 symptom had the same value, the symptom used for analysis was based on the following order of rank: pain>numbness>tingling>discomfort.
Time Frame: From baseline (Day 10 to Day 25 of screening period) to the end of the efficacy follow-up (Day 8 to Day 21).
Population: The ITT-To-Treat (ITT) population, defined as all randomized patients who initiated (received) study drug infusion.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
Number analyzed (Participants) | 97 | 99
Score on a scale | -2.13 [-2.51 to -1.75] | -2.19 [-2.57 to -1.82]

3. Secondary Outcome: Weekly Total Duration of Symptomatic RP Attacks.
Description: The weekly duration is calculated as the average duration of a systematic RP attack times weekly frequency, as registered in electronic diary.
  The baseline weekly duration was calculated as the average duration of a systematic RP attack times weekly frequency during the 10- to 25-day baseline electronic diary completion period.
  The end of the efficacy follow-up weekly duration of symptomatic RP attacks is calculated as the average duration of a systematic RP attack times weekly frequency during Days 8 to 21, inclusive.
Time Frame: From baseline (Day 10 to Day 25 of screening period) to the end of the efficacy follow-up (Day 8 to Day 21).
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
Number analyzed (Participants) | 97 | 99
Minutes | -321.04 [-385.03 to -257.05] | -326.48 [-389.53 to -263.44]

4. Secondary Outcome: Percentage of Responders
Description: The responders are defined as participants that have at least 50% reduction in weekly total duration of symptomatic RP attacks and at least 50% reduction in overall severity from baseline.
  Duration of symptomatic RP attacks and severity of attacks are obtained from electronic diary.
Time Frame: From baseline (Day 10 to Day 25 of screening period) to the end of the efficacy follow-up (Day 8 to Day 21).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
Number analyzed (Participants) | 97 | 99
Participants | 33 | 33

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected during the full study period from the signing of the ICF until the last study visit, Visit 9, at day 35 (+7 days).
Description: For this study, hypotension will be considered an adverse event of special interest (AESI).
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/97 | 1/99
Other Adverse Events (participants affected / at risk) | 78/97 | 99/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=97) | Iloprost Injection, for Intravenous Use (N=99)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=97) | Iloprost Injection, for Intravenous Use (N=99)
Headache (Nervous system disorders) | 38 (82) | 85 (271)
Dizziness (Nervous system disorders) | 10 (14) | 10 (16)
Head discomfort (Nervous system disorders) | 5 (11) | 2 (5)
Paraesthesia (Nervous system disorders) | 5 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (30) | 57 (104)
Vomiting (Gastrointestinal disorders) | 5 (5) | 24 (32)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 13 (20)
Fatigue (General disorders) | 9 (11) | 15 (21)
Infusion site pain (General disorders) | 6 (6) | 15 (18)
Infusion site erythema (General disorders) | 4 (4) | 5 (5)
Asthenia (General disorders) | 2 (2) | 5 (5)
Infusion site extravasation (General disorders) | 1 (1) | 6 (6)
Chills (General disorders) | 1 (1) | 5 (7)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4 (7) | 27 (58)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (9)
Skin ulcer (Skin and subcutaneous tissue disorders) | 12 (22) | 11 (16)
Flushing (Vascular disorders) | 7 (21) | 28 (48)
Palpitations (Cardiac disorders) | 5 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT04040322/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT04040322/SAP_001.pdf